CLINICAL TRIAL: NCT05591365
Title: Effects of Exercise Training on Cardiac Parameters in Coronary Artery Disease Patients After Stenting
Brief Title: Exercise Training in Coronary Artery Disease Patients After Stenting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rec/01277 Pakiza Batool
Record Dates: First submitted 2022-03-30; First posted 2022-10-24 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Stent Restenosis; Coronary Artery Disease
Keywords: Coronary artery diseases; Exercise training; Stenting
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured In-patient and Home plan (Experimental): Structured In-patient and Home plan
  Interventions: Other: Structured In-Patient and Home plan
- Conventional therapy (Placebo Comparator): Conventional protocol as per guidelines
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Other: Structured In-Patient and Home plan — A patient education session and a protocol comprise of 3 days. It consists of three different levels having progressive activities. The in-patient protocol will start from the day of the procedure. Each level contains 2 to 6 tasks, performed in sets of 5-10 repetitions 3 times a day. Home plan: Walking 3 days a week starting from normal pace ((RPE: 8-9) for10 minutes and progressively increased intensity and duration over the period of 12 weeks (RPE: 13-14).
  Arms: Structured In-patient and Home plan
Other: Conventional Therapy — In-Patient: Wound care, Bed mobility:
  AROMS (10 Reps*3sets*TD), Breathing Exercise (10 Reps*3sets*TD), Mobilization (Walk as per patient tolerance) Patient Education: To keep the heart healthy Diet Avoid strenuous exercise and lifting heavy objects Avoid valsalva manure, Quit smoking Lower cholesterol levels, Maintain a healthy weight Control other conditions, such as diabetes and high blood pressure Take medications as prescribed by your doctor Get regular exercise: Walking at a normal pace as per tolerance (RPE up to 10)
  Arms: Conventional therapy

SUMMARY:
To determine the effect of exercise training on cardiac outcomes in coronary artery disease patients after Stenting. There is a need to develop strategies, not only to prevent restenosis but also to improve patients' functional status and perception of well-being. In particular, it is not well defined whether exercise training can reduce the restenosis rate and improve the outcome after PCI.

DETAILED DESCRIPTION:
Based on an analysis of literature reviews, psychological symptoms (such as depression and anxiety), angina, vital exhaustion, and dyspnea have been observed to have the most significant influence on the quality of life in people with CAD. Almost half of the patients, after an initial encouraging improvement in functional capacity and quality of life (QOL) after the PCI, deal with recurrent chest pain that requires medical attention, reduces functional capacity, and creates a status of psychological distress.

ELIGIBILITY:
Inclusion Criteria:

* GCS = 15
* Disease chronicity: 1-3 years
* Elective / stenting procedure
* Single or Double vessel stunting
* EF: 35 above

Exclusion Criteria:

* Unwilling to participate in research
* Known cases of Uncontrolled DM or HTN
* Known cases of Cognitive/memory/neurological disorders
* Known cases of any Systemic disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
6 min walk test: Distance (meters) | 12 weeks
  Changes from the baseline,6th week and 12th week, 6 min walk test (6 MWT) was used to measure Functional capacity. It is a sub maximal exercise test which can aid in assessing functional capacity of patients with cardiopulmonary diseases, in this test we find out the maximum distance in meters which an individual covers in 6 min without any support.
Mindfulness | 12 weeks
  Changes from the Baseline,6th week and 12th week, measured through MAAS. The MAAS is a 15-item scale designed to assess a core characteristic of dispositional mindfulness, namely, open or receptive awareness of and attention to what is taking place in the present. The scale shows strong psychometric properties and has been validated with college, community, and cancer patient samples.Higher scores reflect higher levels of dispositional mindfulness
Rate of perceived exertion (RPE) | 12 weeks
  Changes from the Baseline,6th week and 12th week, measured through Borg RPE scale which measures a person's perception of their effort and exertion breathlessness, and fatigue during physical work rating between 6 and 20. The higher the number, the more intense the exercise. An RPE of 6 is often referred to as just above rest, hardly any exertion, while an RPE of 20 is a maximal effort.
Dyspnea | 12 weeks
  Changes From the Baseline,6th week and 12th week, measured through Rose Dyspnea Scale. The scale consists of four items, with scores ranging from 0 to 4, where 0 indicates no dyspnea with activity, and increasing scores indicate greater limitations because of dyspnea.
Mean arterial pressure | 3-5 days
  Changes From the Baseline, measured through cardiac monitor. Normal range is between 70 and 100 mm Hg.
Heart Rate | 3-5 days
  Changes From the Baseline, measured through Cardiac monitor/Pulse-oximeter. Normal Resting Heart rate ranges from 60 to 100 beats per minute.
Respiratory rate | 3-5 days
  Changes From the Baseline, measured through cardiac monitor. Normal Resting Respiratory rate is12 to 20 breaths per minute
Transcutaneous oxygen saturation [SpO2] | 3-5 days
  Changes From the Baseline, measured through Cardiac monitor/Pulse-oximeter. Normal Resting SpO2 ranges 95% or higher.

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MSPT(CPPT), Principal Investigator — Riphah International University
Locations (1):
- Armed forces institute of cardiology, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No